CLINICAL TRIAL: NCT02950870
Title: An Open-Label Study to Evaluate Long-Term Outcomes With Ombitasvir-Paritaprevir-Ritonavir and Dasabuvir With or Without Ribavirin (RBV) in Fertile Women With Genotype 1 and 4 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Efficacy Study to Evaluate the Effect of New Antiviral Drugs on HCV Infection.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Facchinetti Fabio, PRS administrator, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV_AMH_16
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Hepatitis, C Virus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group treated (Experimental): this group will be treated with Ombitasvir-Paritaprevir-Ritonavir (12,5 mg/75 mg/50 mg) and Dasabuvir ( 250 mg) with or without Ribavirina every day , for 12 weeks.
  Interventions: Drug: Ombitasvir-Paritaprevir-Ritonavir; Drug: Dasabuvir; Drug: Ribavirin
- group untreated (No Intervention): Control group

INTERVENTIONS:
Drug: Ombitasvir-Paritaprevir-Ritonavir — The patient will be treated daily with Ombitasvir-Paritaprevir-Ritonavir 25/150/100 mg total dose
  Other Names: Viekirax
  Arms: group treated
Drug: Dasabuvir — The patient will be treated daily with Dasubavir 500 mg total dose
  Other Names: Exvieria
  Arms: group treated
Drug: Ribavirin — Patients will be treated with ribavirin if necessary.
  Other Names: RBV
  Arms: group treated

SUMMARY:
The purpose of this study is to determinate the AMH levels before and after antiviral therapy with Ombitasvir-Paritaprevir-Ritonavir and Dasabuvir in comparison with age-matched HCV-positive women not undergoing antiviral treatment.

DETAILED DESCRIPTION:
The study is interventional, controlled randomized (block 2:1 case: controls) in open label.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 35 years of age at the time of Screening
* Childbearing potential and sexually active with male partner(s) currently using at least one effective method of birth control at the time of screening and two effective methods of birth control while receiving study drugs, starting with Study Day 1 and for 7 months after stopping study drug.
* Females must have negative results for pregnancy tests
* Chronic HCV-infection prior to study enrollment
* Screening laboratory result indicating HCV GT 1b or GT 1a or GT 4 infection.
* Must be able to voluntarily sign and date an informed consent form
* Liver biopsy within 24 months prior to or during screening demonstrating a Metavir score of 2 or less or an Ishak score of 3 or less or Screening FibroScan® result of ≤ 9.6 kPa;

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Positive test result for HBsAg and HIV Ab
* Recent history of drug or alcohol
* HCV genotype performed during screening indicates more than 1 subtype or co-infection with any other genotype.
* Use of medications contraindicated
* Use of known strong inducers of cytochrome P450 3A (CYP3A) or strong inducers of cytochrome P450 2C8 (CYP2C8) or strong inhibitors of CYP2C8
* History of solid organ transplant.
* Confirmed presence of hepatocellular carcinoma
* Current use of any investigational or commercially available anti-HCV agents
* Screening laboratory analyses showing any of the following abnormal laboratory results

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The modification of AMH levels | 48 weeks post treatment
  The primary outcome is to evaluate the modification of AMH levels before and after successful antiviral therapy in comparison with age-matched HCV-positive women not undergoing antiviral treatment is the primary endpoint

SECONDARY OUTCOMES:
Modification of AMH levels | 144 weeks
  Modification of AMH levels before and after successful antiviral therapy
Modification of the Estradiol (E2) levels | 144 weeks
  Modification of the Estradiol (E2) levels before and after successful antiviral therapy in comparison with age-matched HCV-positive women not undergoing antiviral treatment is the primary endpoint
Percentage of participants experiencing miscarriage | 144 weeks
  Percentage of participants experiencing miscarriage during 3 years observation post-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: ERICA VILLA, Prof., Principal Investigator — Gastroenterology Unit
Locations (1):
- Gastroenterology Unit, Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No